CLINICAL TRIAL: NCT03701698
Title: Ruxolitinib and Methylprednisolone As First Line Therapy for Acute Graft Versus Host Disease Following Allogeneic Stem Cell Transplantation
Brief Title: Ruxolitinib and Steroid As First Line Therapy for Acute GVHD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Participants recruitment failure
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Director, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SHSYXY-Ruxo-GVHD-2018001
Record Dates: First submitted 2018-10-08; First posted 2018-10-10 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Acute GVHD
MeSH Terms: interventions — ruxolitinib; Methylprednisolone; Steroids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- combination therapy (Experimental): There is only 1 arm. Combination therapy arm includes ruxolitinib and methylprednisolone.
  1. Methylprednisolone: 2mg/kg/d , iv or iv gtt for at least 1 week, then taper according to the clinical response.
  2. Ruxolitinib oral tablet, 5~10mg bid orally, for at least 28 days.
  Interventions: Drug: Ruxolitinib Oral Tablet; Drug: Methylprednisolone

INTERVENTIONS:
Drug: Ruxolitinib Oral Tablet — Ruxolitinib Oral Tablet （Jakafi）, 5~10mg bid po for at least 28 days.
  Other Names: Jakafi
Drug: Methylprednisolone — Methylprednisolone: 2mg/kg/d , iv or iv gtt, for at least 1 week, then taper accordingly.
  Other Names: steroid

SUMMARY:
The purpose of this study is to evaluate the efficacy of ruxolitinib in combination with methylprednisolone as first line therapy in patients with Grades II to IV acute graft-versus-host disease (GVHD).

DETAILED DESCRIPTION:
Treatment:

Once patients are diagnosed with grade II~IV acute GVHD, the combination therapy should be initiated as soon as possible.

1. Methylprednisolone: 2mg/kg/d, iv or iv gtt, in two or three divided doses. Taper steroid every one or two weeks according to patient's response.
2. Ruxolitinib 5~10mg bid po for at least 28 days. If patient's ANC<0.5×10e9/L or PLT< 20×10e9/L, cease ruxolitinib until recovery of ANC higher than 0.5×10e9/L or PLT higher than 20×10e9/L.

Indication for stopping Ruxolitinib treatment:

1. No response after ruxolitinib treatment for 28 days.
2. Develop life-threatening complication.
3. ANC<0.5×10e9/L or PLT< 20×10e9/L.

Indication for second line acute GVHD treatment:

1. deterioration of acute GVHD in 3 days
2. no response after 7 days
3. no complete remission after 2 weeks.

Suggestions of second line therapy:

Basiliximab 20mg, d1, d4, d8.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with hematological diseases.
2. recipients of allogeneic peripheral blood stem cell transplantation.
3. new onset of grade II~IV acute graft versus host disease within 100 days post-transplantation.

exclusion criteria:

1. recipients of second allogeneic stem cell transplant.
2. acute GVHD induced by donor lymphocyte infusion, interferon.
3. received treatment other than steroid before enrollment.
4. overlap GVHD syndrome.
5. pregnant or breast-feeding women.
6. absolute neutrophil count (ANC) <0.5×10e9/L or platelet count (PLT) < 20×10e9/L
7. non-GVHD related liver dysfunction: glutamic pyruvic transaminase>= 4 times of upper normal limit, direct bilirubin >= 4 times of upper normal limit
8. renal dysfunction: creatinine clearance < 15 mL/min or glomerular filtration rate< 15 mL/min
9. uncontrolled infection
10. human immunodeficiency virus infection
11. active hepatitis b virus, hepatitis C virus infection and need antivirus treatment.
12. relapse of primary malignant hematological diseases, or graft rejection.
13. allergic history to Janus kinase inhibitors.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
overall response rate | 28 days after treatment
  overall response rate of acute GVHD treatment, including complete response rate and partial response rate after combination therapy.

SECONDARY OUTCOMES:
time to response | 28 days after treatment
  days from beginning to the first day of maximum response
reactivation rate of cytomegalovirus | 100 days within transplant
  reactivation rate of cytomegalovirus infection
1 year incidence of chronic GVHD | 1 year within transplant
  incidence of chronic GVHD 1 year after transplant

CONTACTS AND LOCATIONS:
Overall Officials: Xianmin Song, M.D., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China